CLINICAL TRIAL: NCT06378580
Title: The Prognostic Impact of Surufatinib for the Treatment of Advanced Pancreatic Ductal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Luo Cong (Other)
Responsible Party: Sponsor-Investigator, Luo Cong, Director, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Other Study IDs: LGF22H160084; LGF22H160084 (Other Grant/Funding Number: Zhejiang Provincial Basic Public Welfare Research Program)
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surufatinib combine immune checkpoint inhibitor
  Interventions: Drug: Surufatinib combine immune checkpoint inhibitor
- Chemotherapy
  Interventions: Drug: AG/FOLFIRINOX

INTERVENTIONS:
Drug: Surufatinib combine immune checkpoint inhibitor — Before drug use demographics, blood markers, pathology information# and enhanced CT features.
  Chemotherapy regimens that were combined with surufatinib included AG or FOLFIRINOX regimens. The AG regimen consisted of nab-paclitaxel (125 mg/m2) followed by gemcitabine (1000 mg/m2) on days 1 and 8 every 3 weeks. The FOLFIRINOX regimen included oxalip
  Groups: Surufatinib combine immune checkpoint inhibitor
Drug: AG/FOLFIRINOX — Before drug use demographics, blood markers, pathology information# and enhanced CT features.
  The AG regimen consisted of nab-paclitaxel (125 mg/m2) followed by gemcitabine (1000 mg/m2) on days 1 and 8 every 3 weeks. The FOLFIRINOX regimen included oxaliplatin (85 mg/m2), irinotecan (180 mg/m2), leucovorin (400 mg/m2), and 5-fluorouracil (400 mg/m2 bolus, 2400 mg/m2 continuous intravenous infusion for 46 hours) every 14 days. Both the AG and FOLFIRINOX regimens required completion of 6 cycles or until disease progression or unacceptable toxicity.
  Groups: Chemotherapy

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is a highly aggressive tumor with a poor prognosis, despite the emergence of chemotherapies, unmet medical needs and limited treatment options still exist for patients with metastatic PDAC (mPDAC). Surufatinib is a small-molecule tyrosine kinase inhibitor that targets vascular endothelial growth factor (VEGFR) 1, 2, 3, fibroblast growth factor receptor 1 (FGFR1), and colony stimulating factor 1 receptor (CSF-1R), and ex vivo experiments have demonstrated its effect on PC models.

A retrospective analysis of patients with PDAC who underwent surufatinib at Zhejiang Cancer Hospital (Hangzhou,China) from July 2022 to July 2023.The database was extracted from the preoperative demographics, blood markers, and surgical pathology information of patients undergoing surufatinib in the investigators' hospital.

ELIGIBILITY:
Inclusion Criteria:

(i) were over 18 years old; (ii) had a histological diagnosis of pancreatic adenocarcinoma; (iii) had at least one measurable lesion; (iv) had undergone at least two cycles of surufatinib treatment.

Exclusion Criteria:

(i)non-R0 resection; (ii) Combined with other malignant tumors.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients with mPDAC who received the surufatinib regimen treatment between July 2022 and July 2023 at Zhejiang Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Median progression-free survival | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Province Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Xie Q, Shang C, Jiang L, Ding G, Long D, Luo C. The prognostic impact of surufatinib for the treatment of advanced pancreatic ductal adenocarcinoma: a single center real-world retrospective study. Front Oncol. 2025 May 20;15:1574934. doi: 10.3389/fonc.2025.1574934. eCollection 2025. PMID 40463875